CLINICAL TRIAL: NCT02586246
Title: Long-term Treatment Study of CDP870 Self-injection. A Multicenter, Open-label, Long-term Safety Study to Evaluate the Safety and Efficacy of CDP870 Self-injection Administered at a Dose of 200 mg Biweekly for 24 Weeks or Longer in Patients With Active Rheumatoid Arthritis Who Are Participating in the Long-term Treatment Studies (Study 275-08-002 or Study 275-08-004) of CDP870 Administered Concomitantly With or Without Methotrexate (MTX)
Brief Title: Long-term Treatment Study of CDP870 Self-injection in Patients With Active Rheumatoid Arthritis Who Are Participating in the Long-term Treatment Studies (Study 275-08-002 or Study 275-08-004) of CDP870
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1226-CL-A003; 275-10-001 (Other: UCB)
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Active Rheumatoid Arthritis
Keywords: CDP870; Rheumatoid arthritis; Long-term
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDP870 group from Study 275-08-002 (Experimental): Subjects with active rheumatoid arthritis who are participating in Study 275-08-002 of CDP870
  Interventions: Drug: CDP870
- CDP870 group from Study 275-08-004 (Experimental): Subjects with active rheumatoid arthritis who are participating in Study275-08-004 of CDP870
  Interventions: Drug: CDP870

INTERVENTIONS:
Drug: CDP870 — Self-injection

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of CDP870 self-injection administered for 24 weeks or longer in subjects who are participating in the long-term treatment study (Study 275-08-002 or Study 275-08-004) of CDP870 administered concomitantly with or without Methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed the treatment in the parent clinical studies (NCT00851318 and NCT00850343) up to 52 weeks
* Subjects who are willing to undertake self-injection and provide a written consent

Exclusion Criteria:

* Patients with serious adverse events
* Patients who are judged by the investigator/subinvestigator to be ineligible to participation in the study for reasons such as uncooperative attitude or nonadherence to study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects experiencing at least one adverse event or at least one serious adverse event during the study | The dosing was allowed until launch of certolizumab pegol for RA in Japan. The maximum duration on study drug was 116 weeks.
Percentage of subjects who meet the American College of Rheumatology 20% (ACR20) criteria at Week 12 | at Week 12
Percentage of subjects who meet ACR20 criteria at Week 24 | at Week 24
Percentage of subjects who meet the American College of Rheumatology 50% (ACR50) criteria at Week 12 | at Week 12
Percentage of subjects who meet the American College of Rheumatology 50% (ACR50) criteria at Week 24 | at Week 24
Percentage of subjects who meet the American College of Rheumatology 70% (ACR70) criteria at Week 12 | at Week 12
Percentage of subjects who meet the American College of Rheumatology 70% (ACR70) criteria at Week 24 | at Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (15):
- Japan (15):
  - Aichi
  - Fukuoka
  - Gunma
  - Hiroshima
  - Hokkaido
  - Hyōgo
  - Kagawa
  - Kagoshima
  - Kanagawa
  - Kumamoto
  - Nagasaki
  - Ōita
  - Saitama
  - Tokushima
  - Tokyo

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=1226-CL-A003